CLINICAL TRIAL: NCT05803135
Title: Efficacy and Safety of Iguratimod Combined With Tofacitinib in the Treatment of csDMARD-IR Patients With Active Moderate-to-severe Rheumatoid Arthritis： a Prospective, Randomized, Controlled, Multicenter Study
Brief Title: Iguratimod Combined With Tofacitinib in the Treatment of Rheumatoid Arthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NFEC-2022-282
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: prospective, randomized, controlled, multicenter study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double-Blind Iguratimod (Active Comparator): Iguratimod (25mg twice daily) combined with Tofacitinib (5mg twice daily) for 24 weeks (6 months)
  Interventions: Drug: Iguratimod combined with Tofacitinib;
- Double-Blind Placebo (Placebo Comparator): Placebo (25mg twice daily) combined with Tofacitinib (5mg twice daily) for 24 weeks (6 months)
  Interventions: Drug: Iguratimod combined with Tofacitinib;

INTERVENTIONS:
Drug: Iguratimod combined with Tofacitinib; — Iguratimod (taken orally, 25mg, bid, daily) combined with Tofacitinib (taken orally, 5mg, bid, daily); Placebo of Iguratimod (taken orally, 25mg, bid, daily) combined with Tofacitinib (taken orally, 5mg, bid, daily)
  Other Names: Placebo of Iguratimod combined with Tofacitinib

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Iguratimod combined with Tofacitinib in the treatment of csDMARD-IR patients with active moderate-to-severe rheumatoid arthritis

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a 1-week screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be randomized in a double-blind manner (participant and investigator) in a 1:1 ratio to Iguratimod (25mg, twice daily) combined with Tofacitinib (5mg, twice daily) or placebo (25mg, twice daily) combined with Tofacitinib (5mg, twice daily).

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the following inclusion criteria will be eligible to participate in the study:

1. Male or female aged 18-65 years old;
2. Weight not less than 40kg;
3. Since the diagnosis of RA, the course of disease was ≥6 months;
4. Patients who meet RA standards in 1987 and 2010 ;
5. RA patients with moderate to high disease activity (DAS28 > 3.2) at the time of screening;
6. Active RA (≥6 joints swelling [66 joints count]; ≥Tenderness of 6 joints [68 joint counts]; ESR>28 mm/h or C-reactive protein (CRP) >1.0 mg/dL);
7. Poor response or intolerance to at least one DMARD, including csDMARDs, bDMARDs, but not tsDMARDs;
8. Previous use of any JAK inhibitor was discontinued for six months before enrollment;
9. For patients who have used DMARDs, the washout criteria must be met;
10. Written informed consent;

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study:

* Pregnant or lactating women;
* Platelet count < 10^9/L, or white blood cell < 3*10^9/L, or absolute neutrophil count < 1.2*10^9/L, or Hemoglobin < 9 g/dL or hematocrit <30%;
* According to Cockcroft-Gault, the glomerular filtration rate was ≤40 ml/min.
* ALT>1.5×ULN, AST>1.5×ULN, Cr>135umol/L;
* Subjects with serious cardiovascular, renal, hematologic or endocrine diseases;
* A history of autoimmune rheumatic diseases other than Sjogren's syndrome;
* Subjects with uncontrolled infection;
* Subjects receiving live vaccines within 6 weeks prior to study entry;
* history of alcohol or drug abuse and abstinence for less than 6 months prior to the first use of the study drug;
* Subjects participating in other clinical study within 3 months prior to study entry;
* Have a history of malignant tumor;
* History of recurrent herpes zoster, diffuse herpes zoster;
* People who are allergic to any of the study drugs;
* Other conditions in which the investigator deemed the patient inappropriate for trial entry;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-03-31 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who achieve clinical remission at week 24 using European League Against Rheumatism (EULAR) response criteria DAS28 | week 24
  The proportion of patients with DAS28-CRP<2.6 at the end of 24 weeks was compared between the two groups. The DAS28 is a composite score derived from 4 of these measures，that is the count of tender joint count（TJC, 0-28）and swollen joint count（SJC, 0-28）, measure C reactive protein (CRP, mg/L) and to make a patient assessment of disease activity.

SECONDARY OUTCOMES:
Percentage of American College of Rheumatology [ACR] 20 Criteria Responders at the end of 24 weeks was compared between the two groups. | week 24
  Percentage of American College of Rheumatology [ACR] 20 Criteria Responders at the end of 24 weeks was compared between the two groups.
Percentage of American College of Rheumatology [ACR] 50 Criteria Responders at the end of 24 weeks was compared between the two groups. | week 24
  Percentage of American College of Rheumatology [ACR] 50 Criteria Responders at the end of 24 weeks was compared between the two groups.
Percentage of American College of Rheumatology [ACR] 70 Criteria Responders at the end of 24 weeks was compared between the two groups. | week 24
  Percentage of American College of Rheumatology [ACR] 70 Criteria Responders at the end of 24 weeks was compared between the two groups.
The change of DAS28 score between the two groups at the end of 24 weeks was compared with the baseline value (week 0) | up to week 24
  The change of DAS28 score between the two groups at the end of 24 weeks was compared with the baseline value (week 0)
The change of Clinical Disease Activity Index (CDAI) score between the two groups at the end of 24 weeks was compared with the baseline value (week 0) | up to week 24
  The CDAI is a composite score derived from these measures，that is the count of tender joint count（TJC, 0-28）, swollen joint count（SJC, 0-28）, Patient global assessment（PGA）and physician global assessment（PHGA）, each of the last two was CDAI score will be calculated with formula CDAI = TJC + SJC + PGA + PHGA. CDAI > 22 is considered high disease activity; 10 <CDAI ≤ 22, moderate disease activity; 2.8 <CDAI ≤10, low disease activity; remission is CDAI score ≤2.8.
The change of Simplified Disease Activity Index (SDAI) score between the two groups at the end of 24 weeks was compared with the baseline value (week 0) | up to week 24
  The SDAI is a composite score derived from these measures，that is the count of tender joint count（TJC, 0-28）, swollen joint count（SJC, 0-28）, C-reactive protein (CRP, mg/L), Patient global assessment（PGA）and physician global assessment（PHGA）, each of the last two was assessed on a visual analog scale ranging from 0-10 cm, with higher scores indicating severe disease. SDAI score will be calculated with formula SDAI = TJC + SJC + PGA+PHGA+ CRP. SDAI score exceeding 26 is considered high disease activity; 11 <SDAI ≤26，moderate disease activity; 3.3 <SDAI ≤11, low disease activity; remission is SDAI score ≤ 3.3.
The percentage of patients who achieve clinical remission at week 12 using European League Against Rheumatism (EULAR) response criteria DAS28 | week 12
  The proportion of patients with DAS28-CRP<2.6 at the end of 12 weeks was compared between the two groups. The DAS28 is a composite score derived from 4 of these measures，that is the count of tender joint count（TJC, 0-28）and swollen joint count（SJC, 0-28）, measure C reactive protein (CRP, mg/L) and to make a patient assessment of disease activity.
The proportion of patients with SDAI≤3.3 at the end of 24 weeks was compared between the two groups. | week 24
  The proportion of patients with SDAI≤3.3 at the end of 24 weeks was compared between the two groups.
The proportion of patients with CDAI≤2.8 at the end of 24 weeks was compared between the two groups. | week 24
  The proportion of patients with CDAI≤2.8 at the end of 24 weeks was compared between the two groups.
The changes of ACPA, RF, serum immunoglobulin (IgG, IgA, IgM) levels between the two groups at the end of 24 weeks were compared with the baseline values (week 0). | up to week 24
  The changes of ACPA, RF, serum immunoglobulin (IgG, IgA, IgM) levels between the two groups at the end of 24 weeks were compared with the baseline values (week 0).
The drug retention rate was compared between the two groups at the end of 12 and 24 weeks. | week 12 and 24
  The drug retention rate was compared between the two groups at the end of 12
The proportion of patients with minimal clinically important difference (MCID) of 0.22 on the Health Assessment Questionnaire Disability Index (HAQ-DI) was compared between the two groups at the end of 24 weeks. | week 24
  The proportion of patients with minimal clinically important difference (MCID) of 0.22 on the Health Assessment Questionnaire Disability Index (HAQ-DI) was compared between the two groups at the end of 24 weeks.

OTHER OUTCOMES:
The change of EULAR Sjögren's Syndrome Discasc Activity Index (ESSDAI) score between the two groups associated with Sjögren's Syndrome (SS) at the end of 24 weeks was compared with the baseline value (week 0) | up to week 24
  The change of EULAR Sjögren's Syndrome Discasc Activity Index (ESSDAI) score between the two groups associated with Sjögren's Syndrome (SS) at the end of 24 weeks was compared with the baseline value (week 0)
The change of EULAR Sjögren's Syndrome Patient-Reported Index (ESSPRI) score between the two groups associated with Sjögren's Syndrome (SS) at the end of 24 weeks was compared with the baseline value (week 0) | up to week 24
  The change of EULAR Sjögren's Syndrome Patient-Reported Index (ESSPRI) score between the two groups associated with Sjögren's Syndrome (SS) at the end of 24 weeks was compared with the baseline value (week 0)
Number of participants with"adverse events (AEs)" | up to week 24
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants with"adverse events (AEs)"i.e. physical exam abnormalities，vital sign abnormalities，laboratory value abnormalities，symptom or disease (new or exacerbated) temporally associated with the use of a medicinal product.

IPD SHARING:
Plan to Share IPD: No